CLINICAL TRIAL: NCT01870817
Title: A Pilot Study Investigating the Effect of Post-operative Home Jejunostomy Feeding on Quality of Life and Nutritional Parameters in Patients With Oesophago-gastric Cancer
Brief Title: Home Jejunostomy Feeding Following Esophagectomy/Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: University of Leicester (Other); University of Sheffield (Other); University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34769; PB-PG-0610-22480 (Other Grant/Funding Number: UK NIHR Research for Patient Benefit); 12447 (Other: UKCRN)
Record Dates: First submitted 2013-05-28; First posted 2013-06-06 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Esophageal Neoplasms
Keywords: Randomized; Jejunostomy; Enteral; Nutrition; Esophagectomy; Gastrectomy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home jejunostomy feeding (Active Comparator): Six weeks of post hospital discharge home enteral feeding
  Interventions: Dietary Supplement: Home jejunostomy feeding
- Control (No Intervention): Standard care

INTERVENTIONS:
Dietary Supplement: Home jejunostomy feeding
  Arms: Home jejunostomy feeding

SUMMARY:
After surgery for oesophageal (gullet) or gastric (stomach) cancer, patients are routinely fed by means of a small feeding tube into the intestine (jejunostomy, JEJ) while they are in hospital. Current practice is to stop feeding once the patient leaves hospital, although the tube is left in place for the first 6 weeks. Most patients lose weight after surgery and have to learn to adjust to new eating habits and behaviours. A few patients have the JEJ feed restarted because of nutritional problems and this requires a further inpatient stay.

It is unknown whether every patient would benefit from this type of feeding at home. Previous studies have only assessed the value of JEJ feeding while patients are still in hospital. There is little known about the benefit of continuing JEJ feeding after discharge from hospital, although home feeding is not uncommon in other patient groups (eg. after a stroke).

The proposed study will provide initial information on patients' well being by measuring quality of life and factors such as change in body weight and dietary intake following a period of home JEJ feeding after surgery. Subjects recruited into the study will be placed, randomly, into a control group who receive current nutritional care (based on dietary advice and oral nutritional supplement drinks) or an intervention group who will receive home JEJ feeding for 6 weeks after hospital discharge, in addition to current treatment.

If subjects in the control group are experiencing problems eating at home, home feeding through the JEJ tube will be started as needed.

The study will also examine how surgery and JEJ feeding at home impact on the patient and carer(s) by means of questionnaires and interviews conducted in the patients' home.

Information obtained will assist in the design of a multicentre study. This intervention is considered important because it has the potential to benefit thousands of patients each year at a modest cost.

ELIGIBILITY:
Inclusion Criteria:

* planned esophagectomy or total gastrectomy for adenocarcinoma or squamous carcinoma
* suitable for home enteral nutrition

Exclusion Criteria:

* inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Participant recruitment and retention rates | 7 months
  This pilot study will inform the design and planning of a larger multi-centre study

SECONDARY OUTCOMES:
Quality of life | Recruitment, 3 wks, 6 wks, 3 months, 6 months after surgery
  Variability in disease specific and generic quality of life measures will be assessed
Nutritional parameters | Recruitment, 3 wks, 6 wks, 3 months, 6 months after surgery
  Absolute body weight
Health economics | 7 months
  Estimates of healthcare costs for the duration of the study will be calculated
Readmission rates | 7 months
  Readmission rate to hospital during the study period
Qualitative analysis | 8 weeks
  Interviews will be conducted with up to 10 participants and their carers & thematic qualitative analysis of interviews performed
Food intake | Recruitment, 3 wks, 6 wks, 3 months, 6 months after surgery
  Self-completed 3 day food diaries will be assessed
Nutritional parameters | Recruitment, 3 wks, 6 wks, 3 months, 6 months after surgery
  Body mass index
Nutritional parameters | Recruitment, 3 wks, 6 wks, 3 months, 6 months after surgery
  Mid arm circumference
Nutritional parameters | Recruitment, 3 wks, 6 wks, 3 months, 6 months after surgery
  Triceps fold thickness
Nutritional parameters | Recruitment, 3 wks, 6 wks, 3 months, 6 months after surgery
  Grip strength

CONTACTS AND LOCATIONS:
Overall Officials: David J Bowrey, MD, Study Director — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Baker ML, Halliday V, Robinson P, Smith K, Bowrey DJ. Nutrient intake and contribution of home enteral nutrition to meeting nutritional requirements after oesophagectomy and total gastrectomy. Eur J Clin Nutr. 2017 Sep;71(9):1121-1128. doi: 10.1038/ejcn.2017.88. Epub 2017 Jun 28. PMID 28656968
- [Derived] Bowrey DJ, Baker M, Halliday V, Thomas AL, Pulikottil-Jacob R, Smith K, Morris T, Ring A. A randomised controlled trial of six weeks of home enteral nutrition versus standard care after oesophagectomy or total gastrectomy for cancer: report on a pilot and feasibility study. Trials. 2015 Nov 21;16:531. doi: 10.1186/s13063-015-1053-y. PMID 26590903
- [Derived] Bowrey DJ, Baker M, Halliday V, Thomas AL, Pulikottil-Jacob R, Smith K. Six weeks of home enteral nutrition versus standard care after esophagectomy or total gastrectomy for cancer: study protocol for a randomized controlled trial. Trials. 2014 May 24;15:187. doi: 10.1186/1745-6215-15-187. PMID 24885032
- See also: Published trial protocol — http://www.trialsjournal.com/content/15/1/187